CLINICAL TRIAL: NCT04169048
Title: Preventing Maltreatment and Promoting Mental Health in Children of Mothers With Borderline Personality Disorder - ProChild
Brief Title: Parenting Skills for Mothers With Borderline Personality Disorder (BPD)
Acronym: ProChild
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Freie Universität Berlin (Other)
Collaborators: Ruhr University of Bochum (Other); University of Bremen (Other)
Responsible Party: Principal Investigator, Babette Renneberg, Professor of Clinical Psychology, Freie Universität Berlin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RenRos02
Record Dates: First submitted 2019-10-24; First posted 2019-11-19 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Borderline Personality Disorder; Mothers
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Intervention Model Description: randomized controlled trial with intervention group and waiting group (treatment as usual)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intervention group (BPD) (Experimental): Participants (N=60) receive the weekly conducted intervention (group training for mothers with BPD) over the period of 12 weeks (12 sessions). Assessments of each participant: T0 (pre-intervention), T1 (post-intervention) and follow-up (6 months after T1).
  Interventions: Behavioral: Group training for mothers with Borderline Personality Disorder
- waiting control group (BPD) (No Intervention): Members of this group (N=60) receive no intervention but treatment as usual (TAU). After completing all assessment points (T0, T1, T2), they can receive the intervention of the intervention group (group training).
- clinical control group (AD/MDD) (No Intervention): Mothers with anxiety and/or depression (N=60) receive no intervention. Assessment point only T0.
- healthy control group (No Intervention): Mothers with no actual mental disorder (N=60) receive no intervention.# Assessment points T0, T1, T2.

INTERVENTIONS:
Behavioral: Group training for mothers with Borderline Personality Disorder — The group programme is designed to teach mothers with BPD parenting skills and to reduce dysfunctional parenting attitudes and strategies. The components are: childrens basics needs, mindfulness, stress and stress reduction, dealing with conflicts, dealing with emotions, dysfunctional attitudes, physical contact, parenting rules, self care.
  Arms: Intervention group (BPD)

SUMMARY:
The first disorder-specific parenting training program for mothers with Borderline Personality Disorder (M-BPD) is evaluated in a randomized controlled trial.

The training program is expected to have positive effects on parenting behavior, decrease the risk of maltreatment of the child, and improve emotion regulation in mothers at post treatment and at 6-month follow-up compared to a control group (treatment as usual; TAU).

Additionally, disorder-specific aspects of dysfunctional parenting behavior as well as BPD-specific aspects of child maltreatment are compared to a clinical control group (mothers with anxiety and/or depression, M-AD/D) and a healthy control group (M-CON).

To assess the differential development of parenting, the risk of maltreatment and emotion dysregulation in untreated M-BPD are compared to M-CON. The investigators expect the difference to increase over time, indicating a worsening in BPD parenting.

ELIGIBILITY:
Inclusion criteria for mothers with BPD:

1. diagnosed with BPD (assessed via SCID-PD)
2. running or completed therapy for BPD symptoms
3. child between 6 months and 6 years
4. living with child or regular (weekly) contact

Exclusion criteria for the mothers with BPD

1. Acute child endangerment
2. maternal acute suicidality
3. maternal psychotic symptoms (assessed via SCID-CV)
4. maternal acute alcohol or drug dependency (assessed via SCID-CV)
5. maternal diagnosed intellectual disability.

Inclusion criteria for mothers with depression and/or anxiety disorders:

1. diagnosed with acute affective or anxiety disorder (assessed via SCID-CV)
2. child between 6 months and 6 years
3. living with child or regular (weekly) contact

Exclusion criteria for mothers with depression and/or anxiety disorders:

1. Acute child endangerment
2. maternal acute suicidality
3. maternal psychotic symptoms (assessed via SCID-CV)
4. maternal acute alcohol or drug dependency (assessed via SCID-CV)
5. maternal diagnosed intellectual disability
6. lifetime diagnosis of BPD (assessed via SCID-PD)

Inclusion criteria for healthy control group:

1. child between 6 months and 6 years
2. living with child or regular (weekly) contact

Exclusion criteria for the healthy control group:

1. Acute child endangerment
2. maternal acute suicidality
3. maternal psychotic symptoms (assessed via SCID-CV)
4. maternal acute alcohol or drug dependency (assessed via SCID-CV)
5. maternal diagnosed intellectual disability.
6. lifetime diagnosis of BPD (assessed via SCID-PD)
7. any acute mental disorder (assessed via SCID-CV)
8. current psychotherapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2020-02-04 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Change in dysfunctional discipline practices | day 0 (before treatment), week 12 (after treatment), month 9 (6 months after second assessment)
  Parenting Scale (Arnold, O'Leary, Wolff & Acker, 1993; german version: Erziehungsfragebogen-Kurzform, EFB-K; Miller, 2001). Questionniare measuring dysfunctional discipline practices in parents. Mean values range between 1-7 with higher values indicating more negative parenting strategies.
Change in positive and dysfunctional parenting strategies | day 0 (before treatment), week 12 (after treatment), month 9 (6 months after second assessment)
  Alabama Parenting Questionnaire (Frick, 1991; German DEAPQ-EL-GS; Reichle & Franiek, 2007). The questionnaire assesses several parenting strategies with 7 subscales (positive parenting, responsible parenting, parental Involvement, poor monitoring/supervision, inconsistent discipline, corporal punishment, powerful implementation). Range 6-30, with higher values indicating more of the respective parenting strategy
Change in child rearing competence | day 0 (before treatment), week 12 (after treatment), month 9 (6 months after second assessment)
  Parenting Sense of Competence Scale (PSOC, Gibeau- Wallston & Wandersman, 1978; German FKE; Miller, 2001). The PSOC measures how parents perceive their child rearing competence. Range 0-96 with higher values indicating higher sense of competence.
Change in parental stress | day 0 (before treatment), week 12 (after treatment), month 9 (6 months after second assessment)
  Parental Stress Index (PSI, Abidin, 1995; German EBI; Tröster, 2010). The PSI is a dimensional rating of parental stress. Range 48 - 240 with higher values indicating higher stress.
Change in physical and psychological aggression towards child | day 0 (before treatment), week 12 (after treatment), month 9 (6 months after second assessment)
  Conflict Tactic Scale - Parent Child (CTS-PC; Strauss, 1998). The CTSPC measures the extent to which a parent has carried out specific acts of physical and psychological aggression. Range 0-300 with higher values indicating higher annual frequency
Change in physical abuse potential | day 0 (before treatment), week 12 (after treatment), month 9 (6 months after second assessment)
  Child Abuse Potential Inventory (CAPI, Milner, 1986, German EBSK; Deegener et al., 2009). The CAPI measures physical abuse potential with reference to the individual burden and three validity scales: a lie scale, a random response scale, and an inconsistency scale. t-values are calculated considering all scales.
Change in child neglect | day 0 (before treatment), week 12 (after treatment), month 9 (6 months after second assessment) and for the intervention group after each session.
  Child Neglect Index (CNI; Trocmé, 1996). The CNI measures child neglect, rated by the diagnostician. Range 0-80 with higher values indicating higher neglect.

SECONDARY OUTCOMES:
Change in emotion regulation | day 0 (before treatment), week 12 (after treatment), month 9 (6 months after second assessment)
  Difficulties in Emotion Regulation Scale (DERS; Gratz & Roemer, 2004). Difficulties in emotion regulation are measured with a) awareness and understanding of emotions; (b) acceptance of emotions; (c) the ability to engage in goal-directed behavior, and refrain from impulsive behavior, when experiencing negative emotions; and (d) access to emotion regulation strategies perceived as effective. Range 36 - 180 with higher values indicating more problems in emotion regulation.
Change in mental distress | day 0 (before treatment), week 12 (after treatment), month 9 (6 months after second assessment)
  Brief Symptom Inventory (BSI, Derogatis, 1975; German: Franke, 2000). The BSI measures mental distress. Results are displayed via t-values.
Change in borderline specific thoughts and feelings | day 0 (before treatment), week 12 (after treatment), month 9 (6 months after second assessment)
  Questionnaire of Thoughts and Feelings (QTF, Renneberg et al., 2010). The QTF measures borderline specific thoughts and feelings. Range 1-5 with higher values indicating more BPD-specific thoughts and feelings.

OTHER OUTCOMES:
Negative intervention outcomes | week 12 (after treatment) (intervention group only)
  Questionniare assessing negative intervention outcomes (INEP, Ladwig, Rief, & Nestoriouc, 2014).The INEP measures negative effects of psychotherapy in different areas of life (intrapersonal change, relationships, friendships, family, malpractice, and stigmatization). Range from -3 to +3. Higher values indicating better therapeutic course.
client satisfaction | week 12 (after treatment) (intervention group only)
  Client Satisfaction Questionnaire (CSQ-8, Attkisson & Zwick, 1982; German ZUF-8; Schmidt, Lamprecht & Wittmann, 1989). CSQ-8 measures client satisfaction with intervention. Range 8-32 with higher values indicating greater satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Babette Renneberg, Prof., Principal Investigator — Freie Universität Berlin
Locations (1):
- Freie Universität Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Buck-Hostkotte, S., Renneberg, B. & Rosenbach, C. (2015). Mütter mit Borderline-Persönlichkeitsstörung. Das Trainingsmanual "Borderline und Mutter sein". Weinheim: Beltz.
- [Derived] Rosenbach C, Heinrichs N, Kumsta R, Schneider S, Renneberg B. Study protocol for a multi-center RCT testing a group-based parenting intervention tailored to mothers with borderline personality disorder against a waiting control group (ProChild*-SP1). Trials. 2022 Jul 23;23(1):589. doi: 10.1186/s13063-022-06531-2. PMID 35870944